CLINICAL TRIAL: NCT00700024
Title: The Effect of Testim and Training in a Population Based, Randomized, Placebo-controlled, Double-blinded Study of Hypogonadal Men
Brief Title: Odense Androgen Study - The Effect of Testim and Training in Hypogonadal Men
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Marianne Andersen, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 030
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Hypogonadism; Metabolic Syndrome
Keywords: Body composition; Physical activity; Metabolic syndrome
MeSH Terms: conditions — Hypogonadism; Metabolic Syndrome; Motor Activity | interventions — Testosterone; Testosterone Propionate; Resistance Training; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): testim
  Interventions: Drug: Testim
- 2 (Experimental): placebo
  Interventions: Drug: placebo
- 3 (Experimental): training
  Interventions: Behavioral: Strength training

INTERVENTIONS:
Drug: Testim — 50 mg/dose7day
  Other Names: testosteron
  Arms: 1
Behavioral: Strength training — three times a week
  Other Names: training
  Arms: 3
Drug: placebo — placebo
  Other Names: gel
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of training and testim on Hypogonadism.

DETAILED DESCRIPTION:
The effect of testim and training in hypogonadal men.

ELIGIBILITY:
Inclusion Criteria:

* Male 65-78
* Bioavailable testosterone < 7.3 nmol/L
* Waist > 94 cm

Exclusion Criteria:

* Haematocrit > 0.50
* Known c. prostate or PSA > 3 Myg/L
* Known malignant disease
* Alcohol or drug abuse
* BMI > 40 kg/m2
* Use of 5 alpha reductance inhibitors
* Plan to father children

Ages: 65 Years to 78 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-01 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Lean body mass | january 2008-january 2010

SECONDARY OUTCOMES:
Insulin sensitivity, Visceral fat/liver fat, Body fat, Waist, Physical conditions and physical strengths, Adiponectin, Lipid metabolism, Subjective sensation of energy, Urine cortisol, Sexual function, Serum testosterone | january 2008-january 2010

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, Md, phd, Principal Investigator
Locations (1):
- Odense University Hospital, Odense, Odense, Denmark

REFERENCES:
- [Derived] Kruse R, Petersson SJ, Christensen LL, Kristensen JM, Sabaratnam R, Ortenblad N, Andersen M, Hojlund K. Effect of long-term testosterone therapy on molecular regulators of skeletal muscle mass and fibre-type distribution in aging men with subnormal testosterone. Metabolism. 2020 Nov;112:154347. doi: 10.1016/j.metabol.2020.154347. Epub 2020 Aug 25. PMID 32853647
- [Derived] Jensen RC, Christensen LL, Nielsen J, Schroder HD, Kvorning T, Gejl K, Hojlund K, Glintborg D, Andersen M. Mitochondria, glycogen, and lipid droplets in skeletal muscle during testosterone treatment and strength training: a randomized, double-blinded, placebo-controlled trial. Andrology. 2018 Jul;6(4):547-555. doi: 10.1111/andr.12492. Epub 2018 Apr 15. PMID 29656500
- [Derived] Glintborg D, Christensen LL, Kvorning T, Larsen R, Brixen K, Hougaard DM, Richelsen B, Bruun JM, Andersen M. Strength training and testosterone treatment have opposing effects on migration inhibitor factor levels in ageing men. Mediators Inflamm. 2013;2013:539156. doi: 10.1155/2013/539156. Epub 2013 Sep 8. PMID 24089589
- [Derived] Kvorning T, Christensen LL, Madsen K, Nielsen JL, Gejl KD, Brixen K, Andersen M. Mechanical muscle function and lean body mass during supervised strength training and testosterone therapy in aging men with low-normal testosterone levels. J Am Geriatr Soc. 2013 Jun;61(6):957-962. doi: 10.1111/jgs.12279. Epub 2013 Jun 3. PMID 23730808